CLINICAL TRIAL: NCT03982888
Title: Deep Brain Stimulation for the Treatment of Refractory Repetitive Self-Injurious Behaviour in Children With Autism Spectrum Disorder: A Pilot Project
Brief Title: Deep Brain Stimulation in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, George Ibrahim, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB1000060282
Record Dates: First submitted 2019-06-03; First posted 2019-06-12 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Self-Injurious Behavior
Keywords: deep brain stimulation
MeSH Terms: conditions — Autism Spectrum Disorder; Self-Injurious Behavior | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS Treatment (Experimental): Deep brain stimulation of both limbic and dysfunctional reward processing circuits for treatment of repetitive self injurious behaviours in children with ASD
  Interventions: Procedure: Deep Brain Stimulation; Device: DBS

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Stimulation of the nucleus accumbens via 2 electrodes implanted in the brain per patient to reduce self-injurious behaviours.
Device: DBS — Use of the Medtronic DBS device. DBS device consists of 2 parts:
  1. DBS lead, a thin wire with 2 electrical contacts implanted into pre-determined brain regions, and
  2. Implantable pulse generator, a small device containing the batter and computer source placed under the skin of the chest to generate electrical pulses
  Other Names: Medtronic DBS Therapy (Device # 37601)

SUMMARY:
The purpose of this study is to evaluate the safety and possible effectiveness of deep brain stimulation (DBS) of the nucleus accumbens in children with autism spectrum disorder and treatment-refractory, repetitive self-injurious behavior. Six (6) patients will be recruited and enrolled in this pilot study and study duration for each patient will be one (1) year. All will undergo surgical implantation of the Medtronic DBS system and will receive stimulation of the nucleus accumbens (2 electrodes per patient).This will be an open, non-blinded, non-randomized, pilot, phase I trial.Expected study duration is 36 months.

DETAILED DESCRIPTION:
This is a phase I, non-blinded, non-randomized, pilot trial for safety and efficacy of deep brain stimulation for medically-refractory, repetitive self-injurious behaviours in children with ASD (i.e. secondary stereotypies). The trial will be conducted in compliance with the protocol, GCP and the applicable regulatory requirement(s).

Patients who meet inclusion and exclusion criteria will be identified and recruited the Neurosurgical Clinic at The Hospital for Sick Children. The study will proceed according to the schedule laid out below, and both patients and treating team will be aware of all treatment parameters at all times. Six (6) subjects will be enrolled in this study and study duration for each patient will be one (1) year. Previous phase I trials of DBS in psychiatric and Alzheimer's Disease populations have utilized 6 subjects per surgical target. Such a number is sufficient to demonstrate initial safety, as well as feasibility and clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male patients between age 7-18
* Diagnosis of Autism Spectrum Disorder (as defined by the DSM-5).
* Failure or non eligibility of medical therapy with ongoing repetitive self-injurious behaviours, at 6 months or more after instigation of therapy. Failure is defined as a lack of improvement in self-injurious behaviours, as documented by objective evidence, including caregiver logs or clinician assessment, if the clinician has documented a baseline status prior to instigation of the medical therapy.
* Diagnosis of secondary stereotypies, based on clinical assessment of the treating physicians with evidence of self-injury, documented in the patient records.
* Parents or legal guardians, including caregivers, informed and able to give written consent.
* Able to comply with all testing, follow-ups and study appointments and protocols for 12 months following the end of the duration of the study.

Exclusion Criteria:

* Substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
* Any contraindication to MRI or PET scanning
* Likely to relocate away from the study site or move during the study's one year duration
* Presence of cardiac arrhythmias, or other cardiac, respiratory, renal or endocrine conditions that will result in significant risk from a surgical procedure.
* Pregnancy
* Unable to communicate adequately in English in order to complete the baseline and follow-up questionnaires.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in repetitive behaviour | 1 year
  The Repetitive Behavior Scale-Revised (RBS-R; Bodfish, Symons, Parker & Lewis, 2000) will be used to measure changes in repetitive behaviour pre and post intervention. The following sub-scales will be used:
  * Steretyped behaviour subscale
  * Self-injurious behaviour subscale
  * Compulsive behaviour subscale
  * Ritualistic behaviour subscale
  * Sameness behaviour subscale
  * Restricted behaviour subscale
  All subscales are scored from 0-3 as follows:
  0 = behaviour does not occur
  1. behaviour occurs and is a mild problem
  2. behaviour occurs and is a moderate problem
  3. behaviour occurs and is a severe problem Where a higher number indicates increased repetitive behaviour.
  Subscores are totaled and then an overall score is calculated.
  Measure will be completed at baseline (pre-surgery), weekly from weeks 2-6 post-surgery, bi-weekly from weeks 7-10 post surgery, monthly from weeks 11-51 post-surgery, and 1 year post surgery.
Changes in self-injurious behaviour | 1 year
  The Inventory of Statements about Self-Injury (ISAS; Klonsky & Olino, 2008) will be used to measure changes in self-injurious behaviour pre and post intervention. The scale is scored from 0-2 as follows:
  0= not relevant
  1. somewhat relevant
  2. very relavant Where a higher number indicates increased self-injurious behaviour. Questions are scored and totaled.
  Measure will be completed at baseline (pre-surgery), weekly from weeks 2-6 post-surgery, bi-weekly from weeks 7-10 post surgery, monthly from weeks 11-51 post-surgery, and 1 year post surgery.
Changes in abberant behaviour | 1 year
  The Aberrant Behavior Checklist (Aman, Singh, Stewart & Field, 1985) will be used to measure changes in the extent that abberant behaviour is a problem pre and post intervention. The scale is scored from 0-3 as follows:
  0= not at all a problem
  1. the behaviour is a problem but slight in degree
  2. the problem is moderately serious
  3. the problem is severe in degree Where the higher number indicates the behaviour is problematic. Questions are scored and totaled.
  Measure will be completed at baseline (pre-surgery), weekly from weeks 2-6 post-surgery, bi-weekly from weeks 7-10 post surgery, monthly from weeks 11-51 post-surgery, and 1 year post surgery.
Changes in obsessive-compulsive thoughts | 1 year
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS; Goodman, Price, Rasmussen,1989) will be used to measure changes in the amount of interference of unwanted ideas, images, or impulses pre and post intervention. The scale is scored from 0-4, where 0 represents minimal interference and 4 represents substantial interference. Questions are scored and totaled.
  Measure will be completed at baseline (pre-surgery), weekly from weeks 2-6 post-surgery, bi-weekly from weeks 7-10 post surgery, monthly from weeks 11-51 post-surgery, and 1 year post surgery.
Changes in quality of life | 1 year
  The Paediatric Quality of Life Inventory (PedsQL v. 4.0) will be used to measure changes in self-reported quality of life pre and post intervention. The statements are scored from 0-4 as follows:
  0= it is never a problem
  1 = it is almost never a problem 2= it is sometimes a problem 3 = it is often a problem 4= it is almost always a problem Where a higher score indicates the statement is a problem. All items are scored and totaled.
  Measure will be completed at baseline (pre-surgery), weekly from weeks 2-6 post-surgery, bi-weekly from weeks 7-10 post surgery, monthly from weeks 11-51 post-surgery, and 1 year post surgery.

SECONDARY OUTCOMES:
Changes in physical brain abnormalities | 1 year
  MR images will be analyzed pre and post intervention for the following to assess physical abnormalities of the brain, including type (focal cortical dysplasia, tumor, hippocampal sclerosis, hypothalamic hamartoma, gliosis, brain atrophy), side of abnormalities (left/right/ bilateral), and location (frontal, temporal, sylvian, parietal, occipital, multilobar).
  MRI data will be collected at baseline, 6 weeks post-surgery, and 1 year post-surgery.
Changes in metabolic brain abnormalities | 1 year
  FDG-PET scans will be analyzed to measure changes in neurometabolism pre and post intervention, specifically indications of hypermetabolism in the frontal lobes, hippocampus, and lentiform nucleus.
  FDG-PET data will be collected at baseline, 6 weeks post-surgery, and 1 year post-surgery.
Changes in activity | 1 year
  Changes in activity pre and post intervention will be measured using the Actiwatch Spectrum, Phillips Respironics, Bend, OR. Actigraphy is the continuous measurement of an individual's movement. Actigraph data will be collected at baseline, 6 weeks post-surgery, and 1 year post-surgery. Actigraph data will be analyzed using MATLAB (Mathworks, Natick, MA). Measures analyzed will be maximum and minimum value amplitudes, peak to peak, variance, entropy fast fourier transform, discrete cosine function, z-transform, bispectrum.
Type of adverse events reported in caregiver logs | 1 year
Changes in number of complications pre and post intervention will be compared. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George Ibrahim, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorodetsky C, Mithani K, Breitbart S, Yan H, Zhang K, Gouveia FV, Warsi N, Suresh H, Wong SM, Huber J, Kerr EN, Kulkarni AV, Taylor MJ, P Hagopian L, Fasano A, Ibrahim GM. Deep Brain Stimulation of the Nucleus Accumbens for Severe Self-Injurious Behavior in Children: A Phase I Pilot Trial. Biol Psychiatry. 2025 Jun 15;97(12):1116-1126. doi: 10.1016/j.biopsych.2024.12.001. Epub 2024 Dec 5. PMID 39645140
- [Derived] Yan H, Siegel L, Breitbart S, Gorodetsky C, Fasano A, Rahim A, Loh A, Kulkarni AV, Ibrahim GM. An open-label prospective pilot trial of nucleus accumbens deep brain stimulation for children with autism spectrum disorder and severe, refractory self-injurious behavior: study protocol. Pilot Feasibility Stud. 2022 Feb 2;8(1):24. doi: 10.1186/s40814-022-00988-3. PMID 35109924